CLINICAL TRIAL: NCT03550664
Title: Prediction of the Recovery of Neuromuscular Transmission After Curarization, Pilot Study
Brief Title: Prediction of the Recovery of Neuromuscular Transmission After Curarization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Denis SCHMARTZ, Head of the Anesthesiology department, Brugmann University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CHUB-NMB recovery
Record Dates: First submitted 2018-05-28; First posted 2018-06-08 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Neuromuscular Blockade

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical intervention (Experimental): Patients undergoing a surgical intervention within the CHU Brugmann with utilisation of rocuronium.
  Interventions: Device: Monitoring of neuromuscular transmission

INTERVENTIONS:
Device: Monitoring of neuromuscular transmission — Monitoring of neuromuscular transmission will be done by TOFScan (IdMed, Marseille, France). This device is CE marked, and is used routinely in daily clinical practice. Prior to induction of anesthesia, the TOFScan is placed on a patient's hand and the two stimulation electrodes (ECG electrodes) are placed at the level of the ulnar nerve at the wrist. After induction of anesthesia and before administration of a curare, the TOFScan is calibrated according to the manufacturer's instructions. The TOFScan is placed in automatic mode, it will then automatically adapt its mode of stimulation to the depth of the curarization. The TOFScan measurements will be recorded on a PC connected to the TOFScan.

SUMMARY:
The vast majority of patients receive neuromuscular blockers during surgical procedures, either as a single injection to facilitate intubation or as repeated injections to induce muscle relaxation necessary for surgery. The action of neuromuscular blockers is monitored by measuring the contraction force of the adductor of the thumb after stimulation of the ulnar nerve.Different types of stimulation, such as train-of-four (TOF), post- Tetanus count (PTC), double-burst stimulation (DBS) measure different degrees of curarization.The duration of action of neuromuscular blockers has significant interindividual variability. If the investigators know how to measure the degree of curarization of a patient at a given time, it is difficult to know how long it will take to recover neuromuscular function.

The purpose of this study is to determine if the individual recovery of a patient can be predicted form data obtained at the beginning of his/her recovery curve. The investigators propose to record all neuromuscular transmission monitoring data in 100 patients. From these data, the investigators will try to develop an algorithm that would extrapolate the recovery curve of an isolated patient from the fist neuromuscular monitoring data.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a surgical intervention with rocuronium
* Patients covered by the Belgian social security system

Exclusion Criteria:

* Allergy towards rocuronium
* 20< Body Mass Index <30
* Hepatocellular insufficiency, either clinical or abnormal liver tests
* Renal insufficiency, defined as Modification of diet in renal disease (MDRD) <40ml / min or Cockgroft <50ml / min
* Need to antagonize the curare

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
TOFScan recording | 1 day
  Recordings of the TOFScan device (monitoring of the neuro-muscular transmission) during the entire length of the surgery are automatically stored on PC. This data will be used to conceive a mathematical algorithm predicting the decurarisation curve of an individual patient.

CONTACTS AND LOCATIONS:
Overall Officials: Denis Schmartz, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ortega R, Brull SJ, Prielipp R, Gutierrez A, De La Cruz R, Conley CM. Monitoring Neuromuscular Function. N Engl J Med. 2018 Jan 25;378(4):e6. doi: 10.1056/NEJMvcm1603741. No abstract available. PMID 29365307
- [Background] Heerdt PM, Sunaga H, Savarese JJ. Novel neuromuscular blocking drugs and antagonists. Curr Opin Anaesthesiol. 2015 Aug;28(4):403-10. doi: 10.1097/ACO.0000000000000209. PMID 26087274
- See also: Related Info — https://www.springer.com/gb/book/9783642134760